CLINICAL TRIAL: NCT02999542
Title: The Effect of Intraoperative Music on the Prevalence and Severity of Emergence Delirium in Paediatric Patients: A Randomised Controlled Trial
Brief Title: Effect of Music on Emergence Delirium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Pretoria (Other)
Responsible Party: Principal Investigator, DR. Michelle Olivier, DR, University of Pretoria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 451/2016
Record Dates: First submitted 2016-12-13; First posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Emergence Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Music (Experimental): Children will receive music via headphones
  Interventions: Other: Music
- No music (Experimental): Children will listen to silence via headphones
  Interventions: Other: No music

INTERVENTIONS:
Other: Music — Children will be randomised to receive either music via headphones or silence via headphones
  Arms: Music
Other: No music — Children will be randomised to receive either music via headphones or silence via headphones
  Arms: No music

SUMMARY:
The researchers are conducting a research study to see whether listening to music during an operation will have a positive effect on the way that children wake up from surgery/anaesthetic. It is a common phenomenon where children wake up unhappy, irritated and screaming (known as emergence delirium). Research have shown that music decreases anxiety and pain. The researchers want to see whether music can also influence a child's behaviour after emerging from anaesthesia. In other words whether they will be more calm and cooperative after listening to music while they are asleep during surgery. Should music have a positive effect, anaesthesiologists may use it in future to improve care of patients coming for surgery.

DETAILED DESCRIPTION:
Children coming for certain elective surgeries, where pain has been excluded as a confounding factor, will have headphones placed on their ears after induction of anaesthesia. They will be randomised to two groups, one will receive music and the other just silence. The headphones will be removed just before waking the patient up. In the recovery room the child's behaviour will be observed and will be scored according to a validated score. The two groups will then be compared to see whether music makes a difference to the behaviour after anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2-7 years
* American society of anaesthesiologists class I and II patients
* Child has adequate hearing
* Surgery or procedure under general anaesthesia
* Receiving standardised anaesthetic
* Type of surgeries included: orthopaedic, urological, paediatric surgery and ophthalmology
* Minimum exposure to music must be 15minutes
* Child may not receive any premedication

Exclusion Criteria:

* American society of Anaesthesiologists class 3 and above
* Emergency cases
* Children with hearing problems
* Cognitive impairment

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
The effect of music on the prevalence of emergence delirium in paediatric patients | Up to 12 months

SECONDARY OUTCOMES:
The effect of music therapy on the severity of emergence delirium in paediatric patients. | Up to 12 months

IPD SHARING:
Plan to Share IPD: Undecided